CLINICAL TRIAL: NCT00928577
Title: A Phase IV Prospective Safety Surveillance Cohort Study Of ACAM2000® In Deploying Military Personnel
Brief Title: Safety Surveillance Cohort Study of Vaccinia Vaccine (ACAM2000®)
Status: Completed | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Other Study IDs: H-406-004
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Smallpox
Keywords: Smallpox; Smallpox Vaccine; Vaccinia virus; Military
MeSH Terms: conditions — Smallpox; Vaccinia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ACAM2000 Smallpox Vaccine Group: Participants are vaccinia vaccine-naive and have received ACAM2000 Smallpox vaccine as part of their Service Member readiness process.
- Other vaccinia vaccine Group: Participants did not receive ACAM2000 Smallpox vaccine as part of their Service Member readiness process because they are still protected by previous vaccinia vaccination or are ineligible for current ACAM2000 vaccination either because of recency of prior vaccinia vaccination or for reasons solely attributable to conditions or characteristics of their contacts (such as a healthy soldier who is married to someone with a contraindicated condition).

SUMMARY:
Primary Objectives:

* To compare the rates of myopericarditis (subclinical, suspected, probable, or confirmed) in deploying military subjects who received ACAM2000® vaccine to rates among subjects positioned to deploy who would be personally eligible to receive ACAM2000 vaccine but do not receive ACAM2000 vaccine due to recency of prior vaccination (as determined by DoD healthcare providers) or due to conditions or characteristics of their contacts.
* To identify cases of subclinical myopericarditis in deploying military subjects who received ACAM2000 vaccine.

Secondary Objectives:

* To compare the rates of severe and serious dermatologic adverse events observed in deploying military subjects who received ACAM2000® vaccine to rates among subjects positioned to deploy who would be personally eligible to receive ACAM2000 vaccine but do not receive ACAM2000 vaccine due to recency of prior vaccination (as determined by DoD healthcare providers) or due to conditions or characteristics of their contacts.
* To compare the rates of severe and serious neurological adverse events observed in deploying military subjects who received ACAM2000® vaccine to rates among subjects positioned to deploy who would be personally eligible to receive ACAM2000 vaccine but do not receive ACAM2000 vaccine due to recency of prior vaccination (as determined by DoD healthcare providers) or due to conditions or characteristics of their contacts.
* To compare the rates of adverse events observed in subjects approximately 10 days following their ACAM2000® vaccination to rates among subjects positioned to deploy who would be personally eligible to receive ACAM2000 vaccine but do not receive ACAM2000 vaccine due to recency of prior vaccination (as determined by DoD healthcare providers) or due to conditions or characteristics of their contacts.
* To evaluate potential risk factors associated with the development of confirmed, probable, and/or suspected ACAM2000-associated myopericarditis.

DETAILED DESCRIPTION:
This is a prospective safety surveillance study in a US military Department of Defense (DoD) population. Military subjects either naive to smallpox immunization and have received ACAM2000® vaccine or who have previously been immunized with a vaccinia vaccine, usually Dryvax®, will be enrolled into the study.

No vaccine will be administered as part of this study.

ELIGIBILITY:
Inclusion Criteria :

* Written informed consent obtained prior to the conduct of any study-related procedures.
* Male and Female military personnel positioned for active deployment.
* Participant naïve to previous smallpox vaccination and received the ACAM2000 vaccine (Cohort 1), OR, Participant has not received ACAM2000 vaccine within the prior 3 years, AND is ineligible for current ACAM2000 vaccination either because of recency of prior vaccinia vaccination or for reasons solely attributable to conditions or characteristics of their contacts (such as a healthy soldier who is married to someone with a contraindicated condition) (Cohort 2).

Exclusion Criteria :

* Subjects judged by the investigator as unlikely to understand the scope of the study and/or unlikely to be able to be compliant with the study procedures and visits.
* Participation in any other studies involving investigational or marketed products within 30 days prior to Visit 1.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in Cohort 1 are vaccinia vaccine naive and had received ACAM2000® vaccine as part of their Service Member readiness.
  Participants in Cohort 2 did not receive ACAM2000® vaccine as part of their Service Member readiness process because they are still protected by previous vaccinia vaccination or are ineligible for current ACAM2000 vaccination either because of recency of prior vaccinia vaccination or for reasons solely attributable to conditions or characteristics of their contacts (such as a healthy soldier who is married to someone with a contraindicated condition).
Sampling Method: Non-Probability Sample
Enrollment: 14108 (Actual)
Dates: Start 2008-12; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The percentage and rate per 1,000 of participants with subclinical, suspected, probable, or confirmed myopericarditis following vaccination with either ACAM2000® Smallpox vaccine or other vaccinia vaccine. | Day 10 post-vaccination

SECONDARY OUTCOMES:
Number of participants reporting dermatologic adverse events of rash following vaccination with either ACAM2000 or other vaccinia vaccine | Day 10 post-vaccination
  Dermatologic adverse events of rash are those that meet the following criteria:
  * Serious rashes persisting more than 48 hours that are distant from the vaccination site and
  * associated with systemic symptoms, or
  * involving mucous membranes.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Emergent BioSolutions
Locations (4):
- United States (4):
  - Twentynine Palms, California
  - Fort Campbell North, Kentucky
  - Fort Bliss, Texas
  - Fort Hood, Texas

REFERENCES:
- [Derived] Faix DJ, Gordon DM, Perry LN, Raymond-Loher I, Tati N, Lin G, DiPietro G, Selmani A, Decker MD. Prospective safety surveillance study of ACAM2000 smallpox vaccine in deploying military personnel. Vaccine. 2020 Oct 27;38(46):7323-7330. doi: 10.1016/j.vaccine.2020.09.037. Epub 2020 Sep 20. PMID 32967791